CLINICAL TRIAL: NCT00688012
Title: A Placebo-controlled, Double-blind, Randomized, Single Dose, Dose Escalating Trial in Healthy Men to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SPC3649
Brief Title: Safety Study of SPC3649 in Healthy Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Joan Drejer/Regulatory Manager, Santaris Pharma
Allocation: Randomized | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPC3649-201; EudraCT nummer 2008-001012-20
Record Dates: First submitted 2008-05-07; First posted 2008-06-02 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C
Keywords: antisense; microRna antagonist; anti-miR-122; Safety in healthy volunteers; Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — miravirsen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SPC3649

SUMMARY:
A placebo-controlled, double-blind, randomized, single dose, dose escalating trial in healthy men to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of SPC3649.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteers
* BMI: 19-28 kg/m2
* No clinically significant disease/disorder
* Screening laboratory tests without clinically significant abnormalities, must agree to use condoms during intercourse for one week after study drug infusion
* Following receipt of verbal and written information about the study, the subject must provide signed informed consent before any study related activity is carried out.

Exclusion Criteria:

* Heavy exercise within the past 7 days
* Alcohol intake> 21 units weekly
* Regular smoker
* Received experimental drug within 30 days of study entry
* Planned participation in any experimental study during the study period
* HIV-Ab, HBsAg and/or HCV Ab positive
* History of specific allergy
* Current use of any drug or narcotics.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PhaseOne Trials, Hvidovre University Hospital, Hvidovre, Denmark